CLINICAL TRIAL: NCT06336213
Title: Changes in Antibacterial Therapy Based on Perioperative Dynamics of Presepsin During Reconstructive Thoracic Aorta Surgery
Brief Title: Antibacterial Tactics Based on Presepsin Level in Thoracic Aorta Surgery Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Petrovsky National Research Centre of Surgery (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20240306
Record Dates: First submitted 2024-03-12; First posted 2024-03-28 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Aortic Aneurysm and Dissection; Cardiac Valve Disease; Thoracic Aortic Aneurysm; Thoracic Aortic Dissection
Keywords: biomarkers; presepsin; complications; aortic arch; aorta; aortic aneurysm; ascending aorta; cardiac surgery
MeSH Terms: conditions — Aortic Dissection; Heart Valve Diseases; Aortic Aneurysm, Thoracic; Dissection, Thoracic Aorta; Aortic Aneurysm | interventions — sultamicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ampicillin/sulbactam intervention group (Experimental): If a patient meets dual criteria (presepsin > 519,5 pg/ml at the end of surgery and the absence of presepsin increase after 6 hours after the end of surgery) then switching to ampicillin/sulbactam 3 g every 6 hours at least 72 h after the surgery is done.
  Interventions: Drug: Ampicillin-sulbactam
- Cefazolin (No Intervention): If presepsin < 519,5 pg/ml at the end of surgery, cefazolin 2 g every 6 h at least 72 h p/o is continued further

INTERVENTIONS:
Drug: Ampicillin-sulbactam — If a patient meets dual criteria (presepsin > 519,5 pg/ml at the end of surgery and the absence of presepsin increase after 6 hours after the end of surgery) then switching to ampicillin/sulbactam 3 g every 6 hours at least 72 h after the surgery is done.
  Other Names: sulmacefta, amibactam
  Arms: Ampicillin/sulbactam intervention group

SUMMARY:
According to the literature, presepsin was recommended not only as an effective indicator in the diagnosis of sepsis in intensive care units, but also as a reliable prognostic marker of postoperative inflammatory processes in cardiac surgery. Previous study carried out in Petrovsky NRCS related to biomarkers in cardiac surgery and presepsin in particular showed good sensitivity in infection complications prognosis.

DETAILED DESCRIPTION:
Various biomarkers are being used to improve the quality of prediction models aiming to improve clinical outcomes and reduce mortality in the cardiac surgery patient population. In particular, presepsin and procalcitonin have comparable prognostic value for adverse renal, cardiovascular and respiratory outcomes in cardiac surgery patients. In addition, presepsin has in-hospital, 30-day, and 6-month prognostic mortality rate value and is also highly effective for the early diagnosis of sepsis in patients in the intensive care unit. In the previous study the absence of an increase in the level of presepsin in the first 6 hours after surgery was associated with an increased risk of developing a complicated course of the postoperative period (OR 4.15, 95% CI: 1.83-9.41). The combination of two risk factors - a presepsin level at the end of surgery >519.5 pg/ml and the absence of an increase in the presepsin level in the first 6 hours after surgery was associated with an increased risk of developing a complicated course of the postoperative period (OR 5.80, 95% CI: 2. 19-15.35). The hypothesis of this study suggests that in case of insufficient prevention of infectious complications, based on the dynamics of presepsin, it is permissible to administer the broad-spectrum drug ampicillin/sulbactam 3 g. every 6 hours for at least 72 hours from the date of surgery. It is expected that changes in the tactics of antibacterial therapy will reduce the number of inflammatory complications in patients undergoing surgery on thoracic aorta.

ELIGIBILITY:
Inclusion Criteria:

Thoracic aorta aneurysm/dissection

Exclusion Criteria:

Blood sample hemolysis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-23 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2027-02-15 (Estimated)

PRIMARY OUTCOMES:
Infectious complications rate | up to 10 days
  Postoperative pneumonia, sepsis, wound infection, mediastinitis

SECONDARY OUTCOMES:
Total amount of complicated patients | up to 10 days
  Patients that suffer at least 1 complication in postoperative period
Mortality | up to 10 days
  In-hospital mortality rate
Length of hospital stay | up to 10 days
  Days spent in hospital since admission
Length of ICU stay | up to 10 days
  Hours in ICU after the surgery
Multiorgan failure | up to 10 days
  2 or more organ dysfunction in postoperative period

CONTACTS AND LOCATIONS:
Overall Officials: Boris Akselrod, Professor, Principal Investigator — Petrovsky NRCS
Locations (1):
- Petrovsky Research National Centre of Surgery (Petrovsky NRCS), Moscow, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No